CLINICAL TRIAL: NCT01514123
Title: A Phase I, Open Label, Dose Escalation Study of the VEGF-C Human Monoclonal Antibody VGX-100 Administered by Intravenous Infusion Alone and Co-administered With Bevacizumab in Adult Subjects With Advanced or Metastatic Solid Tumors
Brief Title: Study of VGX-100 Administered Alone and Co-administered With Bevacizumab in Adult Subjects With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Circadian Technologies Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: VGX-100-1001
Record Dates: First submitted 2012-01-12; First posted 2012-01-20 (Estimated); Last update posted 2020-09-17 (Actual); Status verified 2020-09

CONDITIONS: Neoplasms; Cancer
Keywords: VGX-100; Bevacizumab; VEGF-C; First-In-Human; Dose Escalation; Advanced Solid Tumors; Angiogenesis Inhibitors; Angiogenesis Modulating Agents; Pharmacologic Actions; Antibodies, Monoclonal; Phase 1; Oncology; Advanced malignancy
MeSH Terms: conditions — Neoplasms | interventions — Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm A - VGX-100 alone (Experimental): Dose escalation of VGX-100 monotherapy
  Interventions: Drug: VGX-100
- Arm B - VGX-100 plus bevacizumab (Experimental): Dose escalation of VGX-100 in combination with escalating doses of bevacizumab
  Interventions: Drug: VGX-100; Drug: Bevacizumab

INTERVENTIONS:
Drug: VGX-100 — VGX-100 will be administered by IV infusion once every week
Drug: Bevacizumab — Bevacizumab will be administered by IV infusion once every 2 weeks
  Other Names: Avastin
  Arms: Arm B - VGX-100 plus bevacizumab

SUMMARY:
This is a non-randomized, multi-dose, first-in-human, multicenter, two arm (Arm A: VGX-100 alone; Arm B: VGX-100 co-administered with bevacizumab), open label, dose escalation study in subjects with advanced or metastatic solid tumors. The study is aimed at evaluating the safety and establishing the recommended dose of the VEGF-C human monoclonal antibody VGX-100 when administered alone or in combination with bevacizumab.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Provision of written informed consent
* Histologically or cytologically documented advanced or metastatic solid tumor that is refractory to standard treatment, for which no standard therapy is available, or for which the subject refuses standard therapy
* Life expectancy > 3 months in the opinion of the investigator
* ECOG performance status 0 to 1
* Evaluable OR measurable disease by RECIST 1.1 criteria
* Agree to the use of effective contraceptive if either male or female of child bearing potential

Exclusion Criteria:

* Inadequate venous access
* Women who are lactating/breastfeeding
* Women with a positive pregnancy test or who are planning to become pregnant during the duration of the study
* Known to be HIV positive, or have chronic hepatitis B or C
* Major surgical procedure within 6 weeks of Baseline or surgical or other wound that is not fully healed at Baseline
* Untreated or symptomatic brain metastasis, known central nervous system metastasis, or spinal cord compression (except glioblastoma multiforme)
* Mediastinal or cavitated, or lung mass located near, invading or encasing a major blood vessel or airway on imaging
* Squamous cell lung cancer
* History of or known/suspected gastrointestinal perforation
* Hemoptysis of >2.5 mL (half a teaspoon) red blood within 28 days of Screening
* Deep venous thrombosis or history of symptomatic pulmonary thromboembolism within 6 months of Screening
* Gastrointestinal bleeding requiring medical intervention within 28 days of Screening
* Receipt of therapeutic concentrations of warfarin or other anticoagulants within 7 days of Screening
* Receipt of investigational agent(s) for any indication within 28 days of Baseline or 5 half lives, whichever is greater
* Receipt of the following treatments:

  * Traditional cytotoxics, tyrosine kinase inhibitors or other small molecule anti-cancer agents within 21 days
  * Nitrosoureas, mitomycin C, bevacizumab or trastuzumab within 6 weeks
  * Any other therapeutic monoclonal antibodies within 21 days
  * Hormonal therapy (other than gonadal suppression) within 14 days
* Radiotherapy:

  * to >25% bone marrow
  * to brain within 28 days of baseline
  * other than above within 14 days of baseline
* Unstable angina, myocardial infarction, transient ischemic events, or stroke within 24 weeks of Screening
* History of CNS hemorrhage, cerebrovascular hemorrhage, myocardial infarction or reversible posterior leukoencephalopathy syndrome associated with prior anti-VEGF/anti-VEGFR therapy
* Uncontrolled hypertension of ≥ CTCAE Grade 2
* Proteinuria at Baseline of ≥2+ or 1.0g/24 hours
* Prior allergic reaction to a monoclonal antibody

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2011-12-29 (Actual); Primary Completion 2014-02-07 (Actual); Study Completion 2017-11-16 (Actual)

PRIMARY OUTCOMES:
The incidence and severity of adverse events including dose limiting toxicities | Approximately 16 months

SECONDARY OUTCOMES:
Tumor response by RECIST criteria | Approximately 16 months
  Tumor response assessment will be measured by computated tomography (CT) or Magnetic resonance imaging (MRI) every 8 or 12 weeks throughout the study
Pharmacokinetic parameters of VGX-100 alone and co-administered with bevacizumab including Cmax, Cmin, AUC and if feasible half life (t1/2) | 28 days after the last subject in each cohort
Anti-VGX-100 antibody formation | Approximately 16 months
Biomarker levels including VEGF-A, VEGF-C, VEGF-D, soluble VEGFR-2, and soluble VEGFR-3 | Approximately 16 months

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Research, Study Director — Circadian Technologies
Locations (2):
- United States (2):
  - UCLA Hematology-Oncology, Santa Monica, California
  - UT MD Anderson Cancer Center, Houston, Texas

IPD SHARING:
Plan to Share IPD: Undecided